CLINICAL TRIAL: NCT03913819
Title: Prospective Longitudinal Study on the Treatment Outcomes of Various Treatment Modalities Under a Standardized Treatment Protocol in Patients Suffered Substance Abuse Related Voiding Dysfunction
Brief Title: Treatment Outcomes Under a Standardized Treatment Protocol in Patients Suffered Substance Abuse Related Voiding Dysfunction
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Chi Fai, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: CRE-2011.454
Record Dates: First submitted 2019-03-26; First posted 2019-04-12 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Voiding Dysfunction; Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cholinergic Antagonists; Analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- substance abuse group: Patients with voiding dysfunction secondary to substance abuse in a special clinic
  Interventions: Drug: First line treatment: oral NSAID and anticholinergic agents; Drug: Second line treatment: additional treatment for pain control; Drug: Third line treatment: A course of intravesical hyaluronate will be given.; Procedure: Fourth line treatment: surgical intervention

INTERVENTIONS:
Drug: First line treatment: oral NSAID and anticholinergic agents — oral NSAID and anticholinergic agents
Drug: Second line treatment: additional treatment for pain control — Gabapentin, tramadol, Lyrica
Drug: Third line treatment: A course of intravesical hyaluronate will be given. — A course of intravesical hyaluronate will be given.
Procedure: Fourth line treatment: surgical intervention — Consideration of hydrodistention and augmentation cystoplasty

SUMMARY:
With the increase of substance abuse over the world, substance abuse e.g. ketamine and methamphetamine related voiding dysfunction is becoming an important medical problem. However, while the clinical manifestation of the condition is becoming better defined, the underlying pathophysiology is still poorly understood. Moreover, majority of the current treatment is just based on the experience on some small case series and there is no treatment data for larger patient sample or standard recommended treatment in the literature. In order to improve the management of this condition, investigators have formulated a treatment protocol based on the current literatures on the management of voiding dysfunction and also a similar condition, interstitial cystitis / painful-bladder syndrome (IC/PBS). The protocol basically consists of the following modalities:

* Basic information and education on the condition, principle of treatment and psychosocial support.
* First line treatment will include a course of oral anti-inflammatory drugs (for the control of the inflammation process and pain) and anticholinergic agents (for the irritative urinary symptoms).
* If these simple oral medication are found to be not effective, then further treatment will include other oral medications, such as amitriptyline and gabapentin, and some drugs that directly applied into the bladder cavity (hyaluronate) or bladder muscle (botulinum toxin).
* For those patients with intractable symptoms and failed all the above treatments, surgical treatment (hydrodistension, augmentation cystoplasty) will be discussed.

The purpose of this research is to assess the effectiveness of the above treatment protocol in the management of substance induced voiding dysfunction and also assess any possible adverse events related to the usage of the drugs.

DETAILED DESCRIPTION:
With the increase in recreational usage of various soft drugs, such as ketamine, methamphetamine over the world, substance abuse related voiding dysfunction is becoming an important medical problem. However, while the clinical manifestation of the condition is becoming better defined, the underlying pathophysiology is still poorly understood. Moreover, majority of the current treatment is based on the experience on some small case series and there is no treatment data for larger patient sample or standard recommended treatment in the literature. With the rapid increase in patients' demand, there is an urgent need for better clinical study on the effect of various treatment regimes for the condition, to provide more evidence-based recommendation for them. On the other hand, better treatment outcome will also help the rehabilitation of these substance abusers.

However, in Hong Kong, due to the limited funding in the tertiary care health system and the poor social support for the patients, some potential treatment options, including COX II inhibitors, intravesical hyaluronate, and botulinum toxin injection, etc, are not readily available for these patients. Therefore, some patients may receive sub-optimal treatment with more side effects or may have limited access to certain therapeutic options. The patients may have to suffer and this also affects the doctors' experience and hence the formulation of ideal treatment for these patients. If extra or adequate funding is available, it may not only widen the potential treatment options for these patients but also provide more clinical experience and data in guiding the formulation of treatment protocols / recommendation and even guide future research direction.

Therefore, in this proposal, investigators would like to prospectively study the treatment result of various treatment modalities under a standardized treatment protocol. The results will help to evaluate the effectiveness and also tolerability of various proposed treatment options in substance abused related voiding dysfunction. . Because of the certain similarities in the clinical manifestations and pathology of voiding dysfunction and interstitial cystitis / painful-bladder syndrome (IC/PBS), this treatment protocols (referred to later section) will base on standard recommendations of IC/PBS (including the American Urological Guideline) and literature on voiding dysfunction management. For treatment / medications that are not provided in Hospital Authority formulation, investigators will provide to patient if clinically indicated. Currently, because of the insufficient treatment data and also the behavioural characteristics of these substance abusers, it will be difficult or impractical to perform randomized placebo-controlled clinical trials in this area. As a result, a prospective longitudinal study on a standardized treatment protocol is proposed, which will provide some "Real-life practice" information on the management of these patients. The data gathered from this study may also provide basis for future study.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffered substance abuse induced voiding dysfunction

Exclusion Criteria:

* Patient not agreed for consent
* Patient that will not comply to our treatment protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1000 patients suffered from substance abuse induced voiding dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-12-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in total Bladder Capacity after standardized treatment. | Baseline, 4 months, 8 months, 12 months, every 4 months through study completion, and average of 1 year
  Total bladder capacity is assessed by the sum of voided volume and post-voided volume
Change in Pain level after standardized treatment: Pelvic Pain - Urgency Frequency symptom scale | Baseline, 4 months, 8 months, 12 months, every 4 months through study completion, and average of 1 year
  Using the Pelvic Pain - Urgency Frequency symptom scale
Change in Bladder storage function after standardized treatment | Baseline, 4 months, 8 months, 12 months, every 4 months through study completion, and average of 1 year
  Using Overactive Bladder Symptom Score
Change in Bladder voiding function after standardized treatment | Baseline, 4 months, 8 months, 12 months, every 4 months through study completion, and average of 1 year
  Using the International Prostate Symptom Score
Any new Adverse events related to treatment modalities | Baseline, 4 months, 8 months, 12 months, every 4 months through study completion, and average of 1 year
  By patient reporting

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Middela S, Pearce I. Ketamine-induced vesicopathy: a literature review. Int J Clin Pract. 2011 Jan;65(1):27-30. doi: 10.1111/j.1742-1241.2010.02502.x. PMID 21155941
- [Background] Wood D, Cottrell A, Baker SC, Southgate J, Harris M, Fulford S, Woodhouse C, Gillatt D. Recreational ketamine: from pleasure to pain. BJU Int. 2011 Jun;107(12):1881-4. doi: 10.1111/j.1464-410X.2010.10031.x. Epub 2011 Feb 14. PMID 21314885
- [Background] Smith HS. Ketamine-induced urologic insult (KIUI). Pain Physician. 2010 Nov-Dec;13(6):E343-6. No abstract available. PMID 21102971
- [Background] Hanno P, Lin A, Nordling J, Nyberg L, van Ophoven A, Ueda T, Wein A; Bladder Pain Syndrome Committee of the International Consultation on Incontinence. Bladder Pain Syndrome Committee of the International Consultation on Incontinence. Neurourol Urodyn. 2010;29(1):191-8. doi: 10.1002/nau.20847. PMID 20025029
- [Background] Marinkovic SP, Moldwin R, Gillen LM, Stanton SL. The management of interstitial cystitis or painful bladder syndrome in women. BMJ. 2009 Jul 31;339:b2707. doi: 10.1136/bmj.b2707. No abstract available. PMID 19648180
- [Background] Dimitrakov J, Kroenke K, Steers WD, Berde C, Zurakowski D, Freeman MR, Jackson JL. Pharmacologic management of painful bladder syndrome/interstitial cystitis: a systematic review. Arch Intern Med. 2007 Oct 8;167(18):1922-9. doi: 10.1001/archinte.167.18.1922. PMID 17923590